CLINICAL TRIAL: NCT06477263
Title: Preliminary Efficacy and Feasibility of Using NeuroCytotron in the Treatment of Autism Spectrum Disorder: A Pilot Study
Brief Title: NeuroCytotron in the Treatment of Autism Spectrum Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neurocytonix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCX-ASD-01
Record Dates: First submitted 2024-06-05; First posted 2024-06-27 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-08

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm One (Experimental): All participants
  Interventions: Device: Neurocytotron

INTERVENTIONS:
Device: Neurocytotron — Neuronal regeneration treatment

SUMMARY:
Preliminary Efficacy and Feasibility of Using NeuroCytotron in the Treatment of Autism Spectrum Disorder

DETAILED DESCRIPTION:
Experimental, pilot, one-arm, open-label, single-center, 13-month, single-center study to evaluate the effect of NCX neuronal regeneration treatment in subjects with Autism Spectrum Disorder (ASD) to explore the therapeutic effects of NeuroCytonix neuronal regeneration technology on ASD symptoms. Specific objectives include collecting preliminary safety and efficacy data, assessing appropriate dosing, and measuring the impact on participants' quality of life after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects with a confirmed diagnosis of ASD according to DSM-5 criteria.
2. Subjects ≥ 3 and ≤ 50 years.
3. Subjects with ASD severity grade 1 to 3 according to DSM-5 criteria.
4. To have the informed consent of the parents or legal representatives for the subject's participation in the study.
5. Subjects must be physically able and willing to undergo the treatment sessions.
6. Subjects must be medically and psychologically stable to participate in the study.

Exclusion Criteria:

1. Presence of medical conditions that could contraindicate the use of NeuroCytotron DM, such as severe neurological disorders and difficult-to-control epilepsy.

   1. uncontrolled epilepsy is defined as: more than 1 generalized seizure in any month within the 3 months prior to the day 1 visit, or
   2. history of any of the following within 9 months prior to the day 1 visit: prolonged seizures or repetitive seizure activity requiring administration of a rescue benzodiazepine (oral, rectal, etc.) more than once a month, seizures lasting more than 10 minutes, status epilepticus or epilepsy with autonomic involvement.
2. Concurrent participation in other therapies or interventions for autism during the study period.
3. Logistical or situational limitations that prevent regular attendance at treatment sessions.
4. History of significant adverse reactions to similar treatments or involving the use of anesthesia.
5. Presence of serious behavioral problems or aggression that may affect the safety of the subject or staff during treatment sessions.
6. Current or recent (previous 14 days) history of clinically significant bacterial, fungal, viral or mycobacterial infection.
7. Subjects with magnetic implants, pacemakers, claustrophobia or any other condition that prevents them from entering or remaining in the DM NeuroCytotron.

Ages: 3 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-03-06 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Autism Diagnostic Observation Schedule-Second Edition scale scores | Through study completion, an average of 1 year
  * Variables related to social communication, such as quality of social interaction, emotional reciprocity, and verbal and nonverbal communication.
  * Variables related to repetitive and stereotyped behavior, such as repetitive motor movements and restricted interests or behaviors.
  * Autism Diagnostic Observation Schedule-Second Edition total score as a global measure of Autism Spectrum Disorder symptoms.
  The Autism Diagnostic Observation Schedule-Second Edition scores range from 0 to 24, where higher scores indicate a greater severity of Autism Spectrum Disorder symptoms
Changes in Adaptive Behavioral Assessment System scores | Through study completion, an average of 1 year
  * Variables related to adaptive skills in areas such as communication, daily living, personal autonomy and social skills.
  * Total adaptive skills scores to assess overall functioning in different adaptive domains.
  The Autism Diagnostic Observation Schedule-Second Edition scores range from 0 to 24, where higher scores indicate a greater severity of Autism Spectrum Disorder symptoms
  The Adaptive Behavioral Assessment System scores range from 40 to 160, where higher scores indicate better adaptive functioning
Changes in Childhood Autism Rating Scale scores | Through study completion, an average of 1 year
  * Variables related to the severity of ASD symptoms, including aspects such as social relationship, communication, stereotyped behavior and eye contact.
  * Childhood Autism Rating Scale total score as a global measure of Autism Spectrum Disorder symptom severity.
  The Childhood Autism Rating Scale scores range from 15 to 60, where higher scores indicate a greater severity of autism symptoms
Changes in Gilliam Autism Measurement Scale score | Through study completion, an average of 1 year
  * Variables related to the severity of ASD symptoms, including areas such as social interaction, communication, stereotyped behaviors, and restricted interests.
  * Specific subscales of the Gilliam Autism Measurement Scale that assess different dimensions of Autism Spectrum Disorder symptoms.
  The Gilliam Autism Measurement Scale scores range from 0 to 174, where higher scores indicate a greater severity of autism symptoms
Withdrawal Rate | Through study completion, an average of 1 year
  • To assess the study withdrawal rate to NeuroCytotron treatment to determine the feasibility and acceptability of treatment by subjects and caregivers.
Adherence to Treatment | Through study completion, an average of 1 year
  • To assess the adherence to NeuroCytotron treatment to determine the feasibility and acceptability of treatment by subjects and caregivers.
Treatment Security | Through study completion, an average of 1 year
  • Record any treatment-related adverse events to assess the safety of NeuroCytotron in this subject population.
Change in the number of seizures or epileptic seizures during the study period | Through study completion, an average of 1 year
  • Obtain information on the number of seizures (if any) before and after treatment.
Neurophysiological changes: in functional activity and brain anatomy using Magnetic Resonance Imaging | Through study completion, an average of 1 year
  * Representative, visual, motor, basal ganglia and other modules
  * Total brain volume
  * Frontal and temporal lobe volume
  * Cortical thickness in the frontal lobe
  * Surface area and cortical gyrification and cerebrospinal fluid volume
  * Cerebellum volume
  * Volume of the corpus callosum
  * White matter, hippocampus, amygdala, thalamus, and basal ganglia
  The above describes one assessment where several anatomical regions are imaged via Magnetic Resonance Imaging - sequence T1
Neurophysiological changes: in functional activity and brain anatomy using Diffusion Tensor Imaging | Through study completion, an average of 1 year
  • Diffusion Tensor Imaging data, as an increase in the values of the anisotropy fractions (AF)
Neurophysiological changes: in functional activity and brain anatomy using Electroencephalogram | Through study completion, an average of 1 year
  • Brain activities during resting states.

SECONDARY OUTCOMES:
Changes in comorbid symptoms | Through study completion, an average of 1 year
  Evaluate changes in comorbid symptoms commonly associated with Autism Spectrum Disorder
Changes in sensory processing: hypersensitivity by percentile ranks | Through study completion, an average of 1 year
  Measurement of changes in sensory processing difficulties, including hypersensitivity, using standardized tools such as the sensory profile by means of Percentile ranks and classifications on the Sensory Profile 2, which will be administered at baseline (pre-treatment) and after 28 days of treatment (post-treatment).
  Percentile Ranks: Typical Performance: Scores between the 25th and 75th percentiles. Probable Difference: Scores between the 2nd and 25th percentiles or between the 75th and 98th percentiles. Definite Difference: Scores below the 2nd percentile or above the 98th percentile.
  The scores in each sensory domain and the overall sensory profile will be recorded and analyzed to determine changes in sensory processing difficulties.
Changes in sensory processing: hypersensitivity by classification scores | Through study completion, an average of 1 year
  Measurement of changes in sensory processing difficulties, including hypersensitivity, using standardized tools such as the sensory profile by means of Percentile ranks and classifications on the Sensory Profile 2, which will be administered at baseline (pre-treatment) and after 28 days of treatment (post-treatment).
  Classification Scores: Typical Performance: Indicates that the child's sensory processing is within the expected range for their age. Probable Difference: Suggests that the child's sensory processing is somewhat different from peers, possibly affecting their daily life. Definite Difference: Indicates significant differences in sensory processing that are likely to impact daily functioning.
  The scores in each sensory domain and the overall sensory profile will be recorded and analyzed to determine changes in sensory processing difficulties.
Changes in sensory processing: hyposensitivity by percentile ranks | Through study completion, an average of 1 year
  Measurement of changes in sensory processing difficulties, including hyposensitivity, using standardized tools such as the sensory profile by means of Percentile ranks and classifications on the Sensory Profile 2, which will be administered at baseline (pre-treatment) and after 28 days of treatment (post-treatment).
  Percentile Ranks: Typical Performance: Scores between the 25th and 75th percentiles. Probable Difference: Scores between the 2nd and 25th percentiles or between the 75th and 98th percentiles. Definite Difference: Scores below the 2nd percentile or above the 98th percentile.
  The scores in each sensory domain and the overall sensory profile will be recorded and analyzed to determine changes in sensory processing difficulties.
Changes in sensory processing: hyposensitivity by classification scores | Through study completion, an average of 1 year
  Measurement of changes in sensory processing difficulties, including hyposensitivity, using standardized tools such as the sensory profile by means of Percentile ranks and classifications on the Sensory Profile 2, which will be administered at baseline (pre-treatment) and after 28 days of treatment (post-treatment).
  Classification Scores: Typical Performance: Indicates that the child's sensory processing is within the expected range for their age. Probable Difference: Suggests that the child's sensory processing is somewhat different from peers, possibly affecting their daily life. Definite Difference: Indicates significant differences in sensory processing that are likely to impact daily functioning.
  The scores in each sensory domain and the overall sensory profile will be recorded and analyzed to determine changes in sensory processing difficulties.

CONTACTS AND LOCATIONS:
Overall Officials: J R Trujillo, Study Chair — jrtrujillo@neurocytonix.com; Lorenzo R Morales Mancias, Principal Investigator — NeuroCytonix Mexico
Locations (1):
- NeuroCytonix México, San Pedro Garza García, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No